CLINICAL TRIAL: NCT05685433
Title: A Real World Study of eCoin for Urgency Urinary Incontinence: Post Approval Evaluation (RECIPE)
Acronym: RECIPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-5702
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Overactive Bladder; Urge Incontinence; Incontinence, Urinary; Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- eCoin Tibial Nerve Stimulation (Experimental): Subcutaneous stimulation of the tibial nerve using the eCoin device.
  Interventions: Device: eCoin Tibial Nerve Stimulation

INTERVENTIONS:
Device: eCoin Tibial Nerve Stimulation — Subcutaneous stimulation of the tibial nerve using the eCoin device.

SUMMARY:
A prospective, multicenter, single-arm study to evaluate the safety and effectiveness of the eCoin® implanted tibial nerve stimulator in subjects with urgency urinary incontinence (UUI).

DETAILED DESCRIPTION:
The goal of this prospective, multicenter, single-arm study is to assess the long-term safety and effectiveness of the FDA approved eCoin® implanted tibial nerve stimulator in a real world setting. Eligible subjects having overactive bladder (OAB) with urgency urinary incontinence (UUI) will be implanted with the eCoin® implanted tibial stimulator and complete voiding diaries and questionnaires at follow-up visits through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women and men above 18 years old with gender percentages reflective of disease prevalence in the U.S. population
* Individual with diagnosis of overactive bladder with urgency urinary incontinence.
* Individual has at least one urgency urinary incontinence episode on each of three days as determined on a 3-day voiding diary.
* Individual gives written informed consent.
* Individual is mentally competent and able to understand all study requirements.
* Individual is willing and able to complete a 3-day voiding diary and quality of life questionnaire.
* Individual is without pharmacological treatment of overactive bladder (anticholinergic and β3-adrenoceptor agonists) for 2 weeks prior to baseline or longer if the physician judges that the therapeutic effect is still present.
* Individual is intolerant of or has an inadequate response to any of anticholinergics, β3-adrenoceptor agonists, onabotulinumtoxinA, or who have undergone percutaneous tibial nerve stimulation (PTNS).
* Individual is determined to be a suitable surgical candidate by physician.
* Individual is appropriate for eCoin treatment based on the US FDA-approved IFU requirements.

Exclusion Criteria:

* Individual is not appropriate for eCoin therapy based upon the US FDA-approved IFU requirements.
* Individual has clinically significant bladder outlet obstruction. (Suspected bladder outlet obstruction will be initially assessed by uroflow study with those having a maximum flow rate < 15mL/s requiring additional evaluation.)
* Individual has predominantly stress urinary incontinence (greater than 1/3 of leaks on baseline diary are stress).
* Individual has an active urinary tract infection at time of enrollment.
* Individual has known polyuria.
* Individual has significant lower urinary tract pain or has been diagnosed with interstitial cystitis or bladder pain syndrome.
* Individual has abnormal post void residual (i.e. greater than 200 cc initially and on repeat testing after double voiding)
* Individual has clinically significant urethral stricture disease or bladder neck contracture. (Suspected disease or contracture will be initially assessed by uroflow study with those having a maximum flow rate < 15mL/s requiring additional evaluation.)
* Individual has chronic venous insufficiency with a history of skin change (hyperpigmentation, lipodermatosclerosis, ulceration) in the ankle region.
* Individual has morbid obesity and in the opinion of the investigator is not a good candidate for the study.
* Individual has had diagnosis of bladder, urethral, or prostate cancer.
* Individual has had a prior anti-stress incontinence sling surgery within the last year.
* Individual is pregnant or intends to become pregnant during the study.
* Individual has the presence of urinary fistula, bladder stone, or interstitial cystitis.
* Individual has uncontrolled diabetes mellitus (Hemoglobin A1C>7) or diabetes with significant peripheral complications. (Uncontrolled diabetes will be ruled out by blood test excluding those with Hemoglobin A1C>7).
* Individual has an implantable neurostimulator, pacemaker, or implantable cardiac defibrillator (ICD).
* Individual has been treated with onabotulinumtoxinA in the previous 9 months prior to enrollment, or more time if the principal investigator judges that the therapeutic effect is present.
* Individual has been treated with percutaneous tibial nerve stimulation (PTNS) within the previous 4 weeks prior to enrollment or more time if the principal investigator judges that the therapeutic effect is present.
* Individual is currently using transcutaneous electrical nerve stimulation (TENS) in the pelvic region, back, or legs.
* Individual is aware that he or she will need an MRI scan other than a head/neck/shoulder MRI during the study period.
* Individual has a clotting or bleeding disorder or is using anticoagulant therapies and in the opinion of the investigator is not a good candidate for the study (antiplatelet and anticoagulant therapy may be continued or held at the discretion of the investigator).
* Individual is neutropenic or immune-compromised.
* Individual has had previous surgery and/or significant scarring at the implant location.
* Individual has ongoing dermatologic condition at the implant site, including but not limited to dermatitis and autoimmune disorders.
* Individual has a clinically significant peripheral neuropathy in the lower extremities.
* Individual has neurogenic bladder dysfunction.
* Individual has pitting edema at implant location (≥ 2+ is excluded).
* Individual has inadequate skin integrity or any evidence of an infection or inflammation in either lower leg.
* Individual has varicose veins and is symptomatic.
* Individual has open wounds, trauma, or prior surgery in the lower extremities.
* Individual has arterial disease in the lower extremities.
* Individual has vasculitis in the lower extremities.
* Individual has bladder stones or neoplasia. (Suspected bladder stones or neoplasia will be ruled out with a urine dipstick showing no more than trace blood, and microscopic analysis (which should be done in that case) shows ≥3 PBC's /HPF unless that subject has been worked up and found negative for clinically significant disease such as malignant neoplasm or stones.)
* In the opinion of the investigator, Individual is not a good candidate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Responder Rate | 12 months
  Proportion of subjects achieving at least a 50% improvement in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Safety: 12 months rate of all device or procedure related AEs. | 12 months
  Rate of all device or procedure related AEs.

SECONDARY OUTCOMES:
Responder Rate | 24 months
  Proportion of subjects achieving at least a 50% improvement in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Safety Data | 24 months
  Rate of all device or procedure related AEs through 24 months post activation of eCoin.
Safety data through 7 months post-reimplantation. | 7 months post reimplantation
  Rate of device or procedure-related AEs through 7 months post reimplantation.

OTHER OUTCOMES:
Proportion of responders (50% improvement) after 12, 24, 36, 48, and 60 months of therapy. | 12, 24, 36, 48, and 60 months
  Proportion of subjects achieving at least a 50% improvement in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Proportion of responders (75% improvement) after 12, 24, 36, 48, and 60 months of therapy. | 12, 24, 36, 48, and 60 months
  Proportion of subjects achieving at least a 75% improvement in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Proportion of responders (100% improvement) after 12, 24, 36, 48, and 60 months of therapy. | 12, 24, 36, 48, and 60 months
  Proportion of subjects achieving at least a 100% improvement in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Reduction in the number of urgency urinary incontinence episodes. | 12, 24, 36, 48, and 60 months
  Reduction in the number of urgency urinary incontinence episodes on a 3-day voiding diary.
Reduction in the number of urgency urinary incontinence episodes for subjects with 8+ voids per day at baseline. | 12, 24, 36, 48, and 60 months
  Reduction in the number of urgency urinary incontinence episodes on a 3-day voiding diary for subjects who experience more than 8 voids per day at baseline.
Reduction in urgency episodes. | 12, 24, 36, 48, and 60 months
  Reduction in the number of urgency episodes on a 3-day voiding diary.
Reduction in nocturia episodes | 12, 24, 36, 48, and 60 months
  Reduction in nocturia episodes on a 3-day voiding diary.
Patient reported qualify of life | 12, 24, 36, 48, and 60 months
  Improvement in patient reported qualify of life utilizing the Overactive Bladder Symptom Quality of Life Questionnaire (OABq).
Patient reported overactive bladder condition improvement. | 12, 24, 36, 48, and 60 months
  Improvement in patient reported overactive bladder condition utilizing the Patient Global Impression of Improvement (PGI-I) questionnaire.
Patient reported sexual health. | 12 months
  Assess patient reported sexual health using the PROMIS Sexual Function and Satisfaction survey.
Patient reported satisfaction with eCoin. | 12, 24, 36, 48, and 60 months
  Assess patient-reported satisfaction with eCoin therapy using the custom patient satisfaction rating survey.
Device-related adverse events from implantation. | 12, 24, 36, 48, and 60 months
  Rate of device-related adverse events from implantation.
Procedure-related adverse events from implantation. | 12, 24, 36, 48, and 60 months
  Rate of procedure-related adverse events from implantation.
Procedure-related adverse events due to suture technique | 12, 24, 36, 48, and 60 months
  Rate of procedure-related adverse events occurring as a result of inappropriate suture technique.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Urology Centers of Alabama, Homewood, Alabama
  - USA Health, Mobile, Alabama
  - Arkansas Urology, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - AIR Research, Los Angeles, California
  - Stanford Health, Stanford, California
  - Urological Research Network Corp, Hialeah, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - The Iowa Clinic, Ankeny, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc, Kansas City, Kansas
  - Cypress Medical Research, Wichita, Kansas
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Minnesota Urology, Woodbury, Minnesota
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Weill Cornell Medicine: Department of Urology, New York, New York
  - The Oregon Clinic, Portland, Oregon
  - Southern Urogynecology, West Columbia, South Carolina
  - UPNT Research Institute, Arlington, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas